CLINICAL TRIAL: NCT02215408
Title: MEDication Focused Outpatient Care for Underutilization of Secondary Prevention
Acronym: MEDFOCUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Korey Kennelty (Other)
Responsible Party: Sponsor-Investigator, Korey Kennelty, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201309828
Record Dates: First submitted 2014-07-16; First posted 2014-08-13 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Diabetes; Hyperlipidemia; Hypertension; Cardiovascular Disease
Keywords: Diabetes; Hyperlipidemia; Hypertension; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias; Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patient received usual care from the provider in the local clinic.
- CVRS Intervention (Experimental): CVRS pharmacist followed the patient for 12 months in order to decrease the patient's risk of developing cardiovascular disease.
  Interventions: Behavioral: CVRS Intervention

INTERVENTIONS:
Behavioral: CVRS Intervention — A clinical pharmacist working in the University of Iowa CVRS followed each patient for 12 months, working on lifestyle modification and recommending medication changes to the patient's clinical pharmacist in the local clinic.
  Arms: CVRS Intervention

SUMMARY:
The study tested whether a pharmacist-run cardiovascular risk service (CVRS) at the University of Iowa can increase use of national standards of care in clinics

DETAILED DESCRIPTION:
This project conducted a multicenter, cluster-randomized study utilizing a centralized CVRS for medical offices with large geographic, racial and ethnic diversity to determine the extent to which the CVRS model will be implemented. Twenty primary care offices were randomized to either the CVRS arm or a usual care arm, and 18 continued in the study. Each clinic enrolled 20-30 patients per office for a total of 402 subjects, of which 186 represented racial minorities.

Subjects in the intervention arm clinic had regular contact by phone, email or text with a CVRS clinical pharmacist housed at the University of Iowa. The pharmacist communicated with the subject, with the site clinical pharmacist and, as needed, with the site provider to optimize both the subject's pharmaceutical regimen and lifestyle behaviors. The CVRS intervention lasted for 12 months.

A complex algorithm was used to calculate the degree to which the subject's care and medical regimen follows national guidelines for reducing the risk of developing cardiovascular risk.

Post-intervention telephone interviews are being conducted with 20 intervention subjects in order to assess their experience with the intervention and barriers and facilitators to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* English speakers age 55 or greater
* Must have a medical history of at least one of the following:
* Coronary artery disease
* Myocardial infarction
* Stroke
* Transient Ischemic Attack
* Atrial Fibrillation
* Systolic heart failure
* Peripheral vascular disease/claudication
* Carotid artery disease
* Diabetes with either: Low density lipoprotein (LDL) 100 or greater AND/OR systolic blood pressure 140 or higher or diastolic blood pressure 90 or higher

Exclusion Criteria:

* Signs of acute angina, stroke, heart failure or renal failure
* Systolic blood pressure 200 or greater or diastolic blood pressure 115 or greater
* Significant hepatic disease, including: Cirrhosis, Hepatitis B or C infection, Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) 3 times control or higher, or total bilirubin 2.0 mg/dl or higher

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2015-01-20 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
The mean percent of applicable Guideline Advantage standards of care that are met at 12 months | 12 months
  Of the 53 specific standards of care listed in the Guideline Advantage criteria, the mean percent of those standards applicable to each subject that are met at the 12 month time point

SECONDARY OUTCOMES:
The average cost per subject, measured in dollars and cents, of implementing the intervention | 12 months
  The cost per subject will include costs for visits to the primary care physician, the cost of prescribed drugs, and the cost for the time spent by study pharmacists communicating with the patient, creating a care plan, and communicating with the patient's primary care provider.
The percent of intervention group patients who rate the intervention as helpful (versus not helpful) | 24 months
  Of the subset of 20 intervention group patients who are interviewed about the study intervention, the percent who state that the intervention was helpful (versus not helpful).

CONTACTS AND LOCATIONS:
Overall Officials: Barry L. Carter, PharmD, Principal Investigator — University of Iowa; Christopher Coffey, PhD, Principal Investigator — University of Iowa
Locations (18):
- United States (18):
  - University of Florida, Gainesville, Florida
  - University of South Florida, Tampa, Florida
  - Idaho State University, Pocatello, Idaho
  - Midwestern University, Downers Grove, Illinois
  - Genesis Health System, Davenport, Iowa
  - University of Iowa, Iowa City, Iowa
  - Siouxland Medical Education Foundation, Sioux City, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - SUNY-University of Buffalo, Buffalo, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Temple University, Philadelphia, Pennsylvania
  - Texas Tech University Health Science Center, Amarillo, Texas
  - Memorial Hermann Hospital System, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin
  - Wheaton Franciscan Medical Group, Milwaukee, Wisconsin
  - Milwaukee Health Services,Inc., Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) datasets will be created without direct or indirect identifiers and reviewed to make sure that elements cannot be used to potentially identify individual subjects. We will create datasets in transport format and package them along with a copy of the protocol, data dictionaries, and a manual that shows the user how to import the data into their own system. Datasets will include baseline data, interim visit data, ancillary data, procedural based data and outcome data, along with laboratory measurements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 12 months of study completion.
Access Criteria: Requests for data will be evaluated by both the Principal Investigator and the study statistician. Investigators requesting access to the data will be asked to complete a data sharing agreement that provides for: 1) a commitment to using the data only for research purposes and not to attempt to identify any individual participant; 2) a commitment to securing the data using appropriate computer technology; and 3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Background] Carter BL, Coffey CS, Chrischilles EA, Ardery G, Ecklund D, Gryzlak B, Vander Weg MW, James PA, Christensen AJ, Parker CP, Gums T, Finkelstein RJ, Uribe L, Polgreen LA; MEDication Focused Outpatient Care for Underutilization of Secondary Prevention Trial Investigators. A Cluster-Randomized Trial of a Centralized Clinical Pharmacy Cardiovascular Risk Service to Improve Guideline Adherence. Pharmacotherapy. 2015 Jul;35(7):653-62. doi: 10.1002/phar.1603. Epub 2015 Jun 25. PMID 26111939
- [Background] Carter BL, Ardery G. Avoiding Pitfalls With Implementation of Randomized Controlled Multicenter Trials: Strategies to Achieve Milestones. J Am Heart Assoc. 2016 Dec 19;5(12):e004432. doi: 10.1161/JAHA.116.004432. No abstract available. PMID 27993832
- [Derived] Kennelty K, Coffey CS, Ardery G, Uribe L, Yankey J, Ecklund D, James PA, Vander Weg MW, Chrischilles EA, Christensen AJ, Polgreen LA, Gryzlak B, Carter BL. A cluster randomized trial to evaluate a centralized remote clinical pharmacy service in large, health system primary care clinics. J Am Coll Clin Pharm. 2021 Oct;4(10):1287-1299. doi: 10.1002/jac5.1497. Epub 2021 Jul 2. PMID 37265855

DOCUMENTS (1):
  • Study Protocol (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT02215408/Prot_000.pdf